CLINICAL TRIAL: NCT06590857
Title: Phase 1b/2 Open-label Trial of 225Ac-DOTATATE (RYZ101) in Subjects With Estrogen Receptor-positive (ER+), Human Epidermal Growth Factor Receptor 2 (HER2)-Negative, Locally Advanced and Unresectable or Metastatic Breast Cancer Expressing Somatostatin Receptors (SSTRs) and Progressed After Antibody-drug Conjugates and/or Chemotherapy (TRACY-1).
Brief Title: Trial of 225Ac-DOTATATE (RYZ101) in Subjects With ER+, HER2-negative Unresectable or Metastatic Breast Cancer Expressing SSTRs.
Acronym: TRACY-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RayzeBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RYZ101-201
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Breast Cancer; HER2-negative Breast Cancer; ER+ Breast Cancer; Advanced Breast Cancer
Keywords: Actinium; Alpha-Emitter; SSTR+ MBC; ER+, HER2-, MBC; RYZ101; 225Ac; Targeted Radiotherapy; Radiopharmaceutical; SSTR+ ABC; ER+, HER2-, ABC
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): RYZ101 Dose Level -1
  RYZ101 Dose Level 1
  RYZ101 Dose Level 2
  RYZ101 Dose Level 3
  Interventions: Drug: RYZ101
- Expansion (Experimental): RYZ101 RP2D Regimen
  Interventions: Drug: RYZ101

INTERVENTIONS:
Drug: RYZ101 — Ac-225

SUMMARY:
Phase 1b/2 open-label trial of 225Ac-DOTATATE (RYZ101) in subjects with ER+, HER2-negative unresectable or metastatic breast cancer expressing SSTRs.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all the following criteria for enrollment in the study:

* Eastern Cooperative Oncology Group performance status ≤2.
* Histologically confirmed, ER+, HER2-negative, locally advanced and unresectable or metastatic breast cancer not amenable to treatment with curative intent.
* At least one RECIST v1.1-measurable tumor lesion that is SSTR-PET positive (defined as maximum standard uptake value (SUVmax) higher than liver mean standard uptake value (SUVmean) on SSTR-PET imaging) and at least 80% of RECIST v1.1measurable tumor lesions are SSTR-PET positive
* Sufficient renal function, as evidenced by eGFR ≥60 mL/min/1.73m2 calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
* Adequate hematologic and hepatic function

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from the study:

* Prior radiopharmaceutical therapy, including radioembolization.
* Any toxicities from prior treatments that have not recovered to CTCAE Grade ≤1, except for alopecia.
* Significant cardiovascular disease
* Known active uncontrolled or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, spinal cord compression, or leptomeningeal disease.
* History of hypersensitivity or allergy to 225Ac, 68Ga, 64Cu, octreotate, or any of the excipients of DOTATATE imaging agents.
* Prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the study safety or efficacy assessments.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation | 6 weeks of RYZ101 treatment
  Incidence rate of DLTs during the first 6 weeks of RYZ101 treatment
Expansion | Up to approximately 5 years after the last subject has completed RYZ101 treatment
  Overall Response Rate, defined as rate of subjects achieving a Complete Response or Partial Response as determined by BICR using RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Denis Ferreira, MD, Study Director — RayzeBio, Inc.
Locations (23):
- United States (23):
  - Research Facility, Phoenix, Arizona
  - Research Facility, Irvine, California
  - Research Facility, Santa Monica, California
  - Research Facility, Longmont, Colorado
  - Research Facility, Jacksonville, Florida
  - Research Facility, Atlanta, Georgia
  - Research Facility, Indianapolis, Indiana
  - Research Facility, Boston, Massachusetts
  - Research Facility, Detroit, Michigan
  - Research Facility, Rochester, Minnesota
  - Research Facility, St Louis, Missouri
  - Research Facility, Omaha, Nebraska
  - Research Facility, Buffalo, New York
  - Research Facilty, New York, New York
  - Research Facility, New York, New York
  - Research Facility, Cleveland, Ohio
  - Research Facility, Philadelphia, Pennsylvania
  - Research Facility, Pittsburgh, Pennsylvania
  - Research Facility, Dallas, Texas
  - Research Facility, Houston, Texas
  - Research Facilty, Salt Lake City, Utah
  - Research Facility, Norfolk, Virginia
  - Research Facility, Seattle, Washington